CLINICAL TRIAL: NCT02061176
Title: Transanal Haemorrhoidal Dearterialization (THD) Versus Open Haemorrhoidectomy for the Treatment of Haemorrhoids. An Open Prospective Randomized Study.
Brief Title: THD Versus Open Haemorrhoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Per Olov Gunnar Olaison, MD, PhD, Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Holbaek Haemorrhoid Study
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Haemorrhoids; Transanal Haemorrhoidal Dearterialization; Transanal Hemorrhoidal Dearterialisation; Open Haemorrhoidectomy; Open Hemorrhoidectomy
MeSH Terms: conditions — Hemorrhoids | interventions — Hemorrhoidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transanal Haemorrhoidal Dearterialization (Experimental): Patients randomised to Transanal Haemorrhoidal Dearterialization.
  Interventions: Procedure: Transanal Haemorrhoidal Dearterialization
- Open Haemorrhoidectomy (Active Comparator): Patients randomised to Open Haemorrhoidectomy
  Interventions: Procedure: Open Haemorrhoidectomy

INTERVENTIONS:
Procedure: Transanal Haemorrhoidal Dearterialization
  Other Names: Hemorrhoidal Artery Ligation
  Arms: Transanal Haemorrhoidal Dearterialization
Procedure: Open Haemorrhoidectomy
  Other Names: Milligan Morgan; Haemorrhoidectomy
  Arms: Open Haemorrhoidectomy

SUMMARY:
A randomised study comparing Transanal Haemorrhoidal Dearterialization (THD) and Open Haemorrhoidectomy (OH) for the treatment of prolapsing haemorrhoids. The primary aim of the study is to evaluate the long-term effect on haemorrhoidal symptoms one year postoperatively.

Secondary endpoints are postoperative pain, complications, effect on anal continence, recovery and return to normal activity, quality of life and health cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* The patient has Grade III-IV haemorrhoids or Grade II haemorrhoids with bleeding resistant to rubber band ligation or sclerotherapy
* The patient has a Haemorrhoidal Symptom Score of 4 or more
* The patient has an American Society of Anaesthesiologists (ASA) score I-II
* The patient's age is 18-85 years at inclusion
* The patient has had a colonoscopy, sigmoidoscopy or rigid rectoscopy within 3 months before inclusion

Exclusion Criteria:

* The patient has had previous operation for haemorrhoids within the last 2 years
* The patient has had previous operation for anal incontinence
* The patient has an active anal fistula
* The patient has an active anal fissure
* The patient has anal incontinence for solid stools

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Haemorrhoidal Symptoms | 1-year and 5-years postoperatively
  Five questions regarding haemorrhoidal symptoms (pain, bleeding, itching, soiling and prolapse) are used to grade the symptom load. Each symptom is graded from 0-4, giving a total score from 0-20.
  The symptom score is registered preoperatively, 3 and 12 months and 5 years postoperatively.

SECONDARY OUTCOMES:
Postoperative pain | 14 days postoperatively
  Postoperative pain is registered using visual analog scale (VAS), by the hospital staff in the immediate postoperative course during hospital stay and by the patient the first 14 days postoperatively.
Complications | 1-year and 5-years postoperatively
  Early and late complications are registered at 3 and 12 months and 5 years follow up.
Anal continence | 1-year and 5-years postoperatively
  Effect on anal continence is evaluated by Wexner Anal Incontinence Score and Revised Faecal Incotinence Score (RFIS) preoperatively, 3- and 12 months and 5 years postoperatively.
Quality of Life | 1-year and 5-years postoperatively
  QoL is evaluated using Short Health Scale, Short Form(SF)-36 and EQ-5D preoperatively, 1-year and 5-years postoperatively.
Health cost analysis | 1-year and 5-years postoperatively
  Health cost analysis will be based on an estimate of the cost of the operations, recovery of the patients and effect (need for further procedures or medical care).

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Olaison, MD, Ph.D, Principal Investigator — Departement of Surgery, Holbaek County Hospital
Locations (1):
- Departement of Surgery, Holbaek County Hospital., Holbæk, Denmark

REFERENCES:
- [Derived] Rorvik HD, Campos AH, Styr K, Ilum L, McKinstry GK, Brandstrup B, Olaison G. Minimal Open Hemorrhoidectomy Versus Transanal Hemorrhoidal Dearterialization: The Effect on Symptoms: An Open-Label Randomized Controlled Trial. Dis Colon Rectum. 2020 May;63(5):655-667. doi: 10.1097/DCR.0000000000001588. PMID 31996581